CLINICAL TRIAL: NCT03423121
Title: A Phase 1/2 Trial of Tauroursodeoxycholic Acid Supplementation in Progressive MS Patients
Brief Title: A Trial of Bile Acid Supplementation in Patients With Multiple Sclerosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00144766
Record Dates: First submitted 2018-01-12; First posted 2018-02-06 (Actual); Results first posted 2023-05-03 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Progressive Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive | interventions — ursodoxicoltaurine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TUDCA Treatment (Experimental): Tauroursodeoxycholic acid (Taurolite) 250 mg four capsules by mouth, twice daily for 16 weeks.
  Interventions: Drug: Tauroursodeoxycholic Acid
- Placebo oral capsule (Placebo Comparator): Placebo oral capsule four capsules by mouth, twice daily for 16 weeks.
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Tauroursodeoxycholic Acid — Participants will be given 1 gram of Tauroursodeoxycholic acid twice daily in the form of four 250mg capsules.
  Other Names: Taurolite
  Arms: TUDCA Treatment
Drug: Placebo oral capsule — Participants will be given four capsules of the placebo twice daily.
  Arms: Placebo oral capsule

SUMMARY:
This study aims to identify the safety and tolerability of bile acid supplementation in patients with progressive Multiple Sclerosis (MS). Participants will also be assessed for an impact of the bile acid on their immune system and gut microbiome. Half of the participants will receive the bile acid tauroursodeoxycholic acid (TUDCA) and half will receive placebo. The investigators believe participants who take TUDCA will have normalization of blood bile acid levels, a normalization of abnormal immune response and a normalization of the gut microbiome.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Progressive MS based on Lublin Criteria
* Low bile acid levels identified using targeted metabolomics analysis
* On the same therapy for the past 6 months and not expected to switch therapy in the next 6 months
* No relapse in the past 3 months

Exclusion Criteria:

* No previous history of liver disease or cholecystectomy
* No stage IV/V chronic kidney disease or other severe metabolic derangements (e.g. poorly controlled thyroid disease or diabetes)
* BMI < 15 kg/m2 and BMI > 40 kg/m2
* Female patients who are pregnant or nursing, or not willing to use contraception
* Chronic antibiotic use
* Corticosteroid treatment within the past 30 days
* Known history of other neuroinflammatory, neurodegenerative or systemic autoimmune disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2018-06-19 (Actual); Primary Completion 2022-04-28 (Actual); Study Completion 2022-07-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pavan Bhargava, MBBS, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of the 59 people that got enrolled, four (4) were lost to follow-up and did not come for a baseline visit, while one (1) was not eligible based on the screening visit assessments, ending up with 54 people.
Period: Overall Study
Arm/Group | TUDCA Treatment | Placebo Oral Capsule
Started | 28 | 26
Completed | 25 | 20
Not Completed | 3 | 6
Not completed — Lost to Follow-up | 2 | 6
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TUDCA Treatment | Placebo Oral Capsule | Total
Number analyzed (Participants) | 28 | 26 | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (11) | 58 (10) | 57 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 16 | 30
  Male | 14 | 10 | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 28 | 26 | 54
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With at Least One Treatment-related Adverse Event
Description: Safety and tolerability will be assessed based on treatment-related adverse events in the two arms.
Time Frame: 16 weeks
Population: All participants who received at least one dose of the intervention and came back for a follow-up visit.
Measure: Count of Participants; unit: Participants
Arm/Group | TUDCA Treatment | Placebo Oral Capsule
Number analyzed (Participants) | 26 | 21
Participants | 10 | 7

2. Secondary Outcome: Change in Fasting Bile Acid Levels in Plasma
Description: The change of targeted bile acid levels over the course of 16 weeks (duration of the study) is reported.
  Bile acid levels (ng/mL) were log transformed before analysis to approximate normal distribution. Units are log(levels) per 16 weeks. Values are derived from linear mixed-effects models.
Time Frame: Baseline to 16 weeks
Population: All participants who received at least one dose of the intervention and had at least two measurements of bile acid levels in plasma.
Measure: Mean (95% Confidence Interval); unit: log(levels[ng/mL]) per 16 weeks
Arm/Group | TUDCA Treatment | Placebo Oral Capsule
Number analyzed (Participants) | 23 | 20
log(levels[ng/mL]) per 16 weeks
  Chenodeoxycholic Acid | 0.44 [-0.14 to 1.02] | 0.48 [-0.13 to 1.09]
  Cholic Acid | -0.4 [-1.04 to 0.23] | 0.58 [-0.21 to 1.38]
  Deoxycholic Acid | 0.14 [-0.21 to 0.48] | 0.46 [0.13 to 0.8]
  Glycochenodeoxycholic Acid | 0.3 [-0.14 to 0.74] | -0.09 [-0.63 to 0.44]
  Glycocholic Acid | -0.02 [-0.46 to 0.42] | -0.32 [-0.88 to 0.24]
  Glycodeoxycholic Acid | 0.1 [-0.36 to 0.56] | 0.14 [-0.36 to 0.63]
  Glycolithocholic Acid | 0.9 [0.33 to 1.47] | 0.35 [-0.01 to 0.71]
  Glycoursodeoxycholic Acid | 2.3 [1.32 to 3.29] | 0.14 [-0.35 to 0.64]
  Lithocholic Acid | 0.75 [0.28 to 1.22] | 0.2 [-0.12 to 0.51]
  Taurochenodeoxycholic Acid | 0.05 [-0.49 to 0.59] | -0.04 [-0.64 to 0.57]
  Taurocholic Acid | -0.23 [-0.74 to 0.28] | -0.26 [-0.83 to 0.3]
  Taurodeoxycholic Acid | -0.31 [-0.87 to 0.25] | 0.1 [-0.45 to 0.65]
  Taurolithocholic Acid | 0.15 [-0.19 to 0.5] | 0.14 [-0.13 to 0.42]
  Tauroursodeoxycholic Acid | 2.52 [1.3 to 3.73] | -0.22 [-0.52 to 0.07]
  Ursodeoxycholic Acid | 1.89 [0.76 to 3.02] | 0.37 [-0.03 to 0.78]

3. Secondary Outcome: Change in Microbiome Alpha-diversity Measured by Shannon Index at the End of the Study
Description: Change in Shannon index of the gut microbiota between baseline and end of study (16 weeks). Shot-gun metagenomic sequencing in first morning stool specimen was utilized to derive the microbiome composition. Higher values of the index indicate more diversity in the microbial community. The minimum value the Shannon index can take is 0 (no diversity). There is no upper limit to the index.
Time Frame: Baseline to 16 weeks
Population: All participants who received at least one dose of the intervention and returned at least two stool kits were included in the analysis
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | TUDCA Treatment | Placebo Oral Capsule
Number analyzed (Participants) | 21 | 13
score on a scale | -0.15 [-0.47 to 0.18] | 0.06 [-0.3 to 0.41]

4. Secondary Outcome: Change in Flow Cytometric Assessments of Peripheral Blood Mononuclear Cells (PBMCs)
Description: Change in flow cytometric assessments over the course of 16 weeks (duration of the study).
  Cells are expressed as ratios of their parent types. Units reported as change in the ratio per 16 weeks. Values are derived from linear mixed-effects models.
Time Frame: Baseline to 16 weeks
Population: All participants who received at least one dose of the intervention and had at least two blood draws that resulted in PBMC isolation were included in the analysis
Measure: Mean (95% Confidence Interval); unit: parent cell ratio per 16 weeks
Arm/Group | TUDCA Treatment | Placebo Oral Capsule
Number analyzed (Participants) | 23 | 19
parent cell ratio per 16 weeks
  T helper memory cells | -1.34 [-4.63 to 1.96] | 3.05 [-1.88 to 7.98]
  Cytotoxic T memory cells | -1.9 [-5.42 to 1.61] | 2.61 [-2.62 to 7.84]

5. Secondary Outcome: Change in Quality of Life Based on Multiple Sclerosis Quality of Life (MSQOL)-54 Instrument
Description: Change in physical and mental health scores as assessed using the Multiple Sclerosis Quality of Life-54 (MSQOL-54) instrument over the course of 16 weeks (duration of the study). This 54-item instrument generates 12 subscales along with two summary scores, and two additional single-item measures. Two summary scores - physical health and mental health - are derived from a weighted combination of scale scores. Higher scores suggest a better quality of life. Scores can range from 0 to 100.
Time Frame: Baseline to 16 weeks
Population: All participants who received at least one dose of the intervention and completed at least two MSQOL questionnaires were included in the analysis
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | TUDCA Treatment | Placebo Oral Capsule
Number analyzed (Participants) | 19 | 19
score on a scale
  MSQOL - Physical Component | -0.15 [-4.37 to 4.07] | 0.01 [-4.7 to 4.71]
  MSQOL - Mental Component | -0.44 [-4.48 to 3.61] | 4.57 [-0.09 to 9.23]

6. Primary Outcome: Number of Total Treatment-related Adverse Events
Description: Safety and tolerability will be assessed based on treatment-related adverse events in the two arms.
Time Frame: 16 weeks
Population: All participants who received at least one dose of the intervention and came back for a follow-up visit.
Measure: Number; unit: total treatment-related adverse events
Arm/Group | TUDCA Treatment | Placebo Oral Capsule
Number analyzed (Participants) | 26 | 21
total treatment-related adverse events | 11 | 8

7. Primary Outcome: Incidence of Treatment-related Adverse Events (AE)
Description: Safety and tolerability will be assessed based on treatment-related adverse events in the two arms. AE incidence will be measured as total number of events per 1000 exposure years.
Time Frame: 16 weeks
Population: All participants who received at least one dose of the intervention and came back for a follow-up visit.
Measure: Number; unit: total events per 1000 exposure years
Arm/Group | TUDCA Treatment | Placebo Oral Capsule
Number analyzed (Participants) | 26 | 21
total events per 1000 exposure years | 1218 | 1061

ADVERSE EVENTS:
Time Frame: 16 weeks
Description: All participants who received at least one dose of the intervention and had at least one follow-up visit in order to be evaluated for adverse events were considered at risk.
  Two (2) participants in the TUDCA group and five (5) participants in the placebo group were lost to follow-up or withdrew and therefore the number at risk is 26 and 21 for the TUDCA and placebo group, respectively.
Arm/Group | TUDCA Treatment | Placebo Oral Capsule
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/21
Serious Adverse Events (participants affected / at risk) | 1/26 | 0/21
Other Adverse Events (participants affected / at risk) | 9/26 | 7/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TUDCA Treatment (N=26) | Placebo Oral Capsule (N=21)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) — Patient was hospitalized with cholecystitis and bacteremia; received IV antibiotics and improved; discharged after 4 days; underwent cholecystectomy after 2 months
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TUDCA Treatment (N=26) | Placebo Oral Capsule (N=21)
Abdominal cramps (Gastrointestinal disorders) | 2 (2) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 0 (0)
Nausea/Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastroesophageal Reflux (Gastrointestinal disorders) | 2 (2) | 1 (1)
Increased flatulence (Gastrointestinal disorders) | 1 (1) | 1 (1)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Deep Vein Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Facial rash (left) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urinary Tract Infection (Renal and urinary disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-11): https://cdn.clinicaltrials.gov/large-docs/21/NCT03423121/Prot_SAP_000.pdf